CLINICAL TRIAL: NCT05506124
Title: Gynecology Department of Women's Hospital School of Medicine Zhejiang University
Brief Title: Airbag-type Stretchable Electrode Array（ASEA） for Electrical Stimulation in Urinary Incontinence in Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhenwei Xie (Other)
Responsible Party: Sponsor-Investigator, Zhenwei Xie, profressor, Women's Hospital School Of Medicine Zhejiang University
Organization: Women's Hospital School Of Medicine Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZDFY2021-4X102
Record Dates: First submitted 2022-02-22; First posted 2022-08-18 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Urinary Incontinence; Pelvic Floor Muscle Training
Keywords: Urinary incontinence; Pelvic floor muscle training; Pelvic Floor Muscle Electrical Stimulation; Stretchable electronics
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Propose a novel airbag-type stretchable electrode array (ASEA) device for training of the female pelvic floor muscle (PFM) for the treatment of UI
  Interventions: Device: airbag-type stretchable electrode array (ASEA) device
- group 2 (Active Comparator): Propose a two-channel hard electrode device for training of the female pelvic floor muscle (PFM) for the treatment of UI
  Interventions: Device: two-channel hard electrode device

INTERVENTIONS:
Device: airbag-type stretchable electrode array (ASEA) device — Propose a novel airbag-type stretchable electrode array (ASEA) device for electrical stimulation for training of the female pelvic floor muscle (PFM) for the treatment of UI
  Arms: group 1
Device: two-channel hard electrode device — Propose a two-channel hard electrode device for electrical stimulation for training of the female pelvic floor muscle (PFM) for the treatment of UI
  Arms: group 2

SUMMARY:
The prevalence of urinary incontinence increases after the menopause and affects between 38 % and 55 % of women aged over 60 years. Urinary incontinence has a profound impact on quality of life.

Pelvic floor muscle training is the first-line management for urinary incontinence. Electrical stimulation is considered for improving contraction of pelvic floor muscles and aid motivation and adherence to therapy and commonly used in pelvic floor muscle training in clinic therapy. However, the stability and quality of the signals collected by existing stretchable electronics (two-channel hard electrode) are too poor especially when muscle movement is involved, making them inappropriate for aureate pelvic floor muscle training. Here, we propose a physiology-based design method for the stretchable electronics and a novel airbag-type stretchable electrode array (ASEA) device for pelvic floor muscle training.

In this study, the investigators hypothesis that ASEA is effective in controlling UI. A randomized, open, and controlled study will be implemented. "participants with ASEA will be included and be prescribed.

Two-channel hard electrode as electrical stimulation electrode will be used as positive control.The primary efficacy end points is the reduction of symptom scoring and improving of quality-of-life assessment, the frequency of UI at 12th week assessed with bladder diaries and pad testing, and the quality-of-life assessed with incontinence impact questionnaire short form (IIQ-7) and pelvic organ prolapsed-urinary incontinence sexual questionnaire-12(PISQ-12).

The adverse event and medication compliance will be investigated. The aim of this study is to explore the efficacy, safety and therapy of ASEA as electrical stimulation electrode in management of UI. This study will provide new options of electrode for the electrical stimulation in management of UI, which will help improve precision therapy of UI.

DETAILED DESCRIPTION:
The prevalence of the condition increases with age, and it is reported to affect 58%-84% of elderly women. Pelvic floor muscle training is the first-line management for urinary incontinence. Electrical stimulation is considered for improving contraction of pelvic floor muscles and aid motivation and adherence to therapy and commonly used in pelvic floor muscle training in clinic therapy. However, the stability and quality of the existing stretchable electronics are too poor especially when muscle movement is involved, making them inappropriate for high standard clinical treatment. Here, we propose a novel airbag-type stretchable electrode array (ASEA) device for training of the female pelvic floor muscle (PFM) for the treatment of UI. The aim of this study is to explore the efficacy and safety of in management of UI. In this study, the investigators hypothesis that ASEA device therapy is effective in controlling UI. A randomized, open, and controlled study will be implemented. Subjects were recruited in strict accordance the inclusion and exclusion criteria at the outpatient clinic. Patients with UI with Ingelman sundberg graduation (mild, moderate, moderate)≥mild UI will be included. Eligible subjects were randomized according to a computer-generated randomization schedule to to receive two-channel hard electrode or ASEA in a ratio of 1:1. Specific doctors will be designated for the disease diagnosis and treatment.

The investigators were guided by Urinary incontinence and pelvic organ prolapse in women: management (NICE guideline,2019). The primary efficacy end points is the reduction of symptom scoring and improving of quality-of-life assessment. Bladder diaries and pad testing will be to performed to evaluate the frequency and quantify urine loss. The quality-of-life assessed with incontinence impact questionnaire short form (IIQ-7) and pelvic organ prolapsed- urinary incontinence sexual questionnaire-12 (PISQ-12), the higher the score, the greater the impact on the quality of life.

The specification of the CONSORT case report system will be implemented. Sample size assessment according equivalence study. Follow-up and loss cases were strictly controlled. A two-sided test will performed with beta=0.80 and αlpha=0.05. The expected loss rate is calculated at 10%. 29 cases will be enrolled with 58 cases in each group. The study will be accepted regular monitoring and inspection.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of UI
* Have a history of sex
* Menopause≥1 year

Exclusion Criteria:

* Acute reproductive organ inflammation
* With cardiac pacemakers
* Malignant tumors
* History of pelvic radiotherapy
* Pelvic floor surgery≤6 months
* Any disease or symptom that may affect the implementation of the study or the interpretation of the results
* Participate in other clinical trials at the same time

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 58 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of quality of life | Baseline score, Change from Baseline score at 12 weeks
  Use a validated urinary incontinence-specific symptom and quality-of-life questionnaire as follows: Urinary incontinence impact questionnaire IIQ-7, Pelvic organ prolapse / urinary incontinence sexual function questionnaire PISQ-12, Each questionnaire the maximum score is 100 and the minimum score is 0, the higher the score, the worse quality of life.
The change of quantify urine loss | Baseline weight gain, Change from Baseline weight gain at 12 weeks
  The change of urine loss measured by pad test. A pad weight gain≥ 2 g is positive. Mild: 2 g≤ weight gain <5 g; Moderate: 5 g ≤ weight gain < 10 g; Severe: 10 g ≤ weight gain < 50 g; extremely severe Degree: weight gain≥ 50 g. The increasing of weight gain means UI aggravation, while the reduction of weight gain means effective.

SECONDARY OUTCOMES:
The change of symptom scoring | Baseline frequency of symptom scoring, Change from Baseline frequency of symptom scoring at 12 weeks
  Bladder diaries to record the frequency of symptom scoring. The increasing of frequency of symptom scoring means UI aggravation, while the reduction of frequency of symptom scoring means effective.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenwei Xie, MD, Principal Investigator — Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu JM, Vaughan CP, Goode PS, Redden DT, Burgio KL, Richter HE, Markland AD. Prevalence and trends of symptomatic pelvic floor disorders in U.S. women. Obstet Gynecol. 2014 Jan;123(1):141-148. doi: 10.1097/AOG.0000000000000057. PMID 24463674
- [Background] Zuchelo LTS, Bezerra IMP, Da Silva ATM, Gomes JM, Soares Junior JM, Chada Baracat E, de Abreu LC, Sorpreso ICE. Questionnaires to evaluate pelvic floor dysfunction in the postpartum period: a systematic review. Int J Womens Health. 2018 Aug 8;10:409-424. doi: 10.2147/IJWH.S164266. eCollection 2018. PMID 30123009
- [Background] Tinelli A, Malvasi A, Rahimi S, Negro R, Vergara D, Martignago R, Pellegrino M, Cavallotti C. Age-related pelvic floor modifications and prolapse risk factors in postmenopausal women. Menopause. 2010 Jan-Feb;17(1):204-12. doi: 10.1097/gme.0b013e3181b0c2ae. PMID 19629013
- [Background] Koenig I, Luginbuehl H, Radlinger L. Reliability of pelvic floor muscle electromyography tested on healthy women and women with pelvic floor muscle dysfunction. Ann Phys Rehabil Med. 2017 Nov;60(6):382-386. doi: 10.1016/j.rehab.2017.04.002. Epub 2017 Jul 14. PMID 28716538